CLINICAL TRIAL: NCT00003590
Title: Phase II Study of Hydroxyurea for Unresectable Meningioma
Brief Title: S9811 Hydroxyurea in Treating Patients With Unresectable Benign Meningioma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH); Eastern Cooperative Oncology Group (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000066659; S9811 (Other: SWOG); ECOG-S9811 (Other: ECOG); U10CA032102 (NIH)
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Results first posted 2012-02-16 (Estimated); Last update posted 2016-05-20 (Estimated); Status verified 2016-04

CONDITIONS: Adult Meningioma
Keywords: recurrent adult brain tumor; adult grade I meningioma
MeSH Terms: conditions — Meningioma; Brain Neoplasms | interventions — Hydroxyurea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Hydroxyurea (Experimental)
  Interventions: Drug: hydroxyurea

INTERVENTIONS:
Drug: hydroxyurea — 20 mg/kg/day PO

SUMMARY:
RATIONALE: Drugs used in chemotherapy such as hydroxyurea use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: This phase II trial is studying how well hydroxyurea works in treating patients with unresectable benign meningioma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the partial and complete response rates in patients with unresectable benign meningioma treated with hydroxyurea.
* Assess the quantitative and qualitative toxic effects of this drug in this patient population.

OUTLINE: Patients receive oral hydroxyurea twice daily for 2 years in the absence of disease progression or unacceptable toxicity.

Patients are followed at 3 months, 6 months, and then every 6 months for 3 years.

PROJECTED ACCRUAL: A total of 38 patients will be accrued for this study within 13 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed unresectable primary, recurrent, or residual benign meningioma
* Measurable disease by CT scan or MRI
* Must have disease progression within the past 10 years OR progressive neurologic deficit within the past 6 months
* Must have undergone prior radiotherapy with subsequent disease progression OR refused radiotherapy

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* SWOG 0-2

Life expectancy:

* Not specified

Hematopoietic:

* WBC at least 4,000/mm^3
* Platelet count at least lower limit of normal

Hepatic:

* Not specified

Renal:

* Not specified

Other:

* Not pregnant or nursing
* Fertile patients must use effective contraception
* No other malignancy within the past 5 years except adequately treated basal or squamous cell skin cancer, carcinoma in situ of the cervix, or adequately treated stage I or II cancer in complete remission

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No prior cytotoxic chemotherapy for meningioma
* Prior mifepristone allowed
* No other concurrent chemotherapy

Endocrine therapy:

* Concurrent glucocorticoids and hormone replacement therapy allowed if stable dose maintained for at least 72 hours prior to CT scan or MRI
* No concurrent antitumor hormonal therapy

Radiotherapy:

* See Disease Characteristics
* At least 6 months since prior radiotherapy
* No concurrent radiotherapy

Surgery:

* Not specified

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 1998-11; Primary Completion 2008-12 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lode J. Swinnen, MD, Study Chair — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins; Geoffrey R. Barger, MD, Study Chair — Barbara Ann Karmanos Cancer Institute
Locations (133):
- United States (133):
  - Fairbanks Cancer Treatment Center at Fairbanks Memorial Hospital, Fairbanks, Alaska
  - St. Joseph's Hospital and Medical Center, Phoenix, Arizona
  - CCOP - Western Regional, Arizona, Phoenix, Arizona
  - Arkansas Cancer Research Center at University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - University of California Davis Cancer Center, Sacramento, California
  - University of Colorado Cancer Center at University of Colorado Health Sciences Center, Aurora, Colorado
  - St. Anthony Central Hospital, Denver, Colorado
  - Denver Health Medical Center, Denver, Colorado
  - Veterans Affairs Medical Center - Denver, Denver, Colorado
  - Montrose Memorial Hospital Cancer Center, Montrose, Colorado
  - St. Anthony North Hospital, Westminster, Colorado
  - Exempla Lutheran Medical Center, Wheat Ridge, Colorado
  - M.D. Anderson Cancer Center - Orlando, Orlando, Florida
  - North Idaho Cancer Center, Coeur d'Alene, Idaho
  - Rush-Copley Cancer Care Center, Aurora, Illinois
  - St. Joseph Medical Center, Bloomington, Illinois
  - Graham Hospital, Canton, Illinois
  - Memorial Hospital, Carthage, Illinois
  - University of Illinois Medical Center, Chicago, Illinois
  - Veterans Affairs Medical Center - Chicago Westside Hospital, Chicago, Illinois
  - Eureka Hospital, Eureka, Illinois
  - Galesburg Clinic, Galesburg, Illinois
  - Galesburg Cottage Hospital, Galesburg, Illinois
  - InterCommunity Cancer Center of Western Illinois, Galesburg, Illinois
  - Mason District Hospital, Havana, Illinois
  - Hopedale Medical Complex, Hopedale, Illinois
  - Joliet Oncology Hematology Associates, Limited - West, Joliet, Illinois
  - Kewanee Hospital, Kewanee, Illinois
  - McDonough District Hospital, Macomb, Illinois
  - Edward Hospital Cancer Center, Naperville, Illinois
  - BroMenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center, Normal, Illinois
  - Community Hospital of Ottawa, Ottawa, Illinois
  - Oncology Hematology Associates of Central Illinois - Ottawa, Ottawa, Illinois
  - Cancer Treatment Center at Pekin Hospital, Pekin, Illinois
  - Proctor Hospital, Peoria, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - Oncology/Hematology Associates of Central Illinois, P.C., Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF St. Francis Medical Center, Peoria, Illinois
  - Illinois Valley Community Hospital, Peru, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - St. Margaret's Hospital, Spring Valley, Illinois
  - Valley Cancer Center, Spring Valley, Illinois
  - Carle Cancer Center at Carle Foundation Hospital, Urbana, Illinois
  - Carle Clinic Association, Urbana, Illinois
  - Saint Anthony Memorial Health Centers, Michigan City, Indiana
  - Siouxland Hematology-Oncology Associates, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, P.A. - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Kingman, Kingman, Kansas
  - Southwest Medical Center, Liberal, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Cancer Center of Kansas - Ottawa, Ottawa, Kansas
  - Cancer Center of Kansas, P.A. - Parsons, Parsons, Kansas
  - Pratt Cancer Center of Kansas, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates in Womens Health, Wichita, Kansas
  - Cancer Center of Kansas, P.A. - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Mary Bird Perkins Cancer Center - Baton Rouge, Baton Rouge, Louisiana
  - Baton Rouge General Regional Cancer Center, Baton Rouge, Louisiana
  - Cancer Center at Medical Center of Louisiana - New Orleans, New Orleans, Louisiana
  - DeCesaris Cancer Institute at Anne Arundel Medical Center, Annapolis, Maryland
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Josephine Ford Cancer Center at Henry Ford Health System, Detroit, Michigan
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Mercy and Unity Cancer Center at Mercy and Unity Hospitals, Fridley, Minnesota
  - Virginia Piper Cancer Institute at Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hubert H. Humphrey Cancer Center at North Memorial Medical Center, Robbinsdale, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Clinic, Saint Louis Park, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Veterans Affairs Medical Center - Kansas City, Kansas City, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Riverside Methodist Hospital Cancer Care, Columbus, Ohio
  - Mount Carmel West Hospital, Columbus, Ohio
  - Doctors Hospital at Ohio Health, Columbus, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Community Oncology Group - Independence, Independence, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Strecker Cancer Center at Marietta Memorial Hospital, Marietta, Ohio
  - Licking Memorial Cancer Care Program at Licking Memorial Hospital, Newark, Ohio
  - Mercy Medical Center Oncology Unit, Springfield, Ohio
  - Community Hospital of Springfield and Clark County, Springfield, Ohio
  - Rose Ramer Cancer Clinic at Anderson Area Medical Center, Anderson, South Carolina
  - CCOP - Greenville, Greenville, South Carolina
  - Sioux Valley Hospital and University of South Dakota Medical Center, Sioux Falls, South Dakota
  - Avera McKennan Hospital and University Health Center, Sioux Falls, South Dakota
  - Medical X-Ray Center, Sioux Falls, South Dakota
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - Wilford Hall Medical Center, Lackland Air Force Base, Texas
  - Center for Cancer Prevention and Care at Scott and White Clinic, Temple, Texas
  - American Fork Hospital, American Fork, Utah
  - Logan Regional Hospital, Logan, Utah
  - Cottonwood Hospital Medical Center, Murray, Utah
  - McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center - Provo, Provo, Utah
  - Huntsman Cancer Institute at University of Utah, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Dixie Regional Medical Center, St. George, Utah
  - Grays Harbor Community Hospital, Aberdeen, Washington
  - Auburn Regional Center for Cancer Care at Auburn Regional Medical Center, Auburn, Washington
  - St. Francis Hospital, Federal Way, Washington
  - Cascade Cancer Center at Evergreen Hospital Medical Center, Kirkland, Washington
  - St. Clare Hospital, Lakewood, Washington
  - Capital Medical Center, Olympia, Washington
  - Providence St. Peter Hospital Regional Cancer Center, Olympia, Washington
  - Olympic Medical Center, Port Angeles, Washington
  - Good Samaritan Cancer Center, Puyallup, Washington
  - Valley Medical Center, Renton, Washington
  - CCOP - Virginia Mason Research Center, Seattle, Washington
  - CCOP - Northwest, Tacoma, Washington
  - St. Joseph Medical Center at Franciscan Health System, Tacoma, Washington
  - Allenmore Hospital, Tacoma, Washington
  - Camden-Clark Memorial Hospital, Parkersburg, West Virginia

REFERENCES:
- [Result] Swinnen LJ, Rankin C, Rushing EJ, et al.: Phase II study of hydroxyurea for unresectable meningioma (Southwest Oncology Group S9811). [Abstract] J Clin Oncol 27 (Suppl 15): A-2063, 2009.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was activated on November 15, 1998 and closed to accrual on June 1, 2005. This was open to all SWOG institutions with IRB approval. Eastern Cooperative Oncology Group (ECOG) joined this trial on May 14, 2004.
Pre-assignment Details: All registered patients were to have eligibility assessed and sign informed consent prior to registration and receipt of protocol therapy.
Groups:
- Hydroxyurea: Only eligible patients were included in the analyses.
  Patients received 20 mg/kg/day taken orally.
Period: Overall Study
Arm/Group | Hydroxyurea
Started | 29
Eligible | 28
Eligible and Began Protocol Therapy | 28
Completed | 7 (Patients were to receive Hydroxyurea up to 2 years in absence of progressive disease.)
Not Completed | 22
Not completed — Ineligible Patient | 1
Not completed — Adverse Event | 7
Not completed — Withdrawal by Subject | 1
Not completed — Lack of Efficacy | 11
Not completed — Death | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | Hydroxyurea
Number analyzed (Participants) | 28
Age, Continuous [Median (Full Range); unit: years] | 62 [24 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Ethnicity was captured at baseline and is reported per NIH/OMB categorization.
  Participants
    Hispanic or Latino | 1
    Not Hispanic or Latino | 27
    Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Race of participant was collected at baseline and is reported per the NIH/OMB categorization.
  Participants
    American Indian or Alaska Native | 0
    Asian | 0
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 0
    White | 28
    More than one race | 0
    Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 28

OUTCOME MEASURES:

1. Primary Outcome: Assess Number of Patients Who Achieve Confirmed and Unconfirmed Complete Response (CR) or Partial Response (PR)
Description: Complete Response (CR)is a complete disappearance of all measurable and evaluable disease. No new lesions, no disease related symptoms, no evidence of non-evaluable disease. Partial Response (PR)is greater than or equal to 50% decrease under baseline in sum of the products of perpendicular diameters of all measurable lesions. No progression of evaluable disease, no new lesions. Confirmation of CR or PR means a repeat scan at least 3 weeks apart documented before progression. No response means that patient did not achieve complete or partial response (either confirmed or unconfirmed).
Time Frame: Patients treated for 2 years or progression. If responding can continue at physician's discretion.
Population: All eligible patients who started treatment were included in assessing response estimates.
Measure: Number; unit: Participants
Groups:
- Hydroxyurea: Patients received 20 mg/kg/day PO.
Arm/Group | Hydroxyurea
Number analyzed (Participants) | 28
Participants
  Complete Response (CR) | 0
  Confirmed Partial Response (PR) | 0
  Unconfirmed Complete Response (UCR) | 0
  Unconfirmed Partial Response (UPR) | 0
  No Response | 28

2. Secondary Outcome: Number of Patients With Gr 3 Through 5 Adverse Events That Are Related to Study Drug
Description: Adverse Events (AEs) are reported by CTC 2.0 terminology. For each patient, worst grade of each event type is reported. Grade 3 - Severe, Grade 4 - Life-threatening, Grade 5 - Fatal
Time Frame: Patients were assessed for adverse events 4 weeks after starting treatment. Assessments for adverse events continued every 3 months for the duration of protocol therapy. On average patients remained on therapy for 8 months
Population: Eligible patients who had received any hydroxyurea were included in the adverse event summaries. Any CTC 2.0 event of Grade 3 (serious), Grade 4 (life threatening) or Grade 5 (fatal) which were deemed to be related to protocol treatment are included.
Measure: Number; unit: Participants with a given type of AE
Arm/Group | Hydroxyurea
Number analyzed (Participants) | 28
Participants with a given type of AE
  Anemia | 1
  Confusion | 1
  Dyspnea | 1
  Fatigue/malaise/lethargy | 1
  Headache | 2
  Hypoxia | 1
  Inner ear-hearing loss | 1
  Leukopenia | 3
  Lymphopenia | 2
  Neutropenia/granulocytopenia | 10
  Respiratory infect w/o neutrop | 1
  Respiratory infection, unk ANC | 1
  Syncope | 1
  Thrombocytopenia | 1

ADVERSE EVENTS:
Time Frame: Patients were assessed for adverse events 4 weeks after starting treatment. Assessments for adverse events continued every 3 months for the duration of protocol therapy. On average patients remained on therapy for 8 months.
Groups:
- Hydroxyurea: Patients received Hydroxyurea (20 mg/kg/day orally) up to 2 years in absence of progressive disease.
Arm/Group | Hydroxyurea
Serious Adverse Events (participants affected / at risk) | 0/28
Other Adverse Events (participants affected / at risk) | 28/28
OTHER ADVERSE EVENTS (reported when occurring in more than 0.05% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Hydroxyurea (N=28)
Anemia (Blood and lymphatic system disorders) | 3
Constipation/bowel obstruction (Gastrointestinal disorders) | 3
Diarrhea without colostomy (Gastrointestinal disorders) | 6
Dyspepsia/heartburn (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 12
Stomatitis/pharyngitis (Gastrointestinal disorders) | 3
Edema (General disorders) | 8
Fatigue/malaise/lethargy (General disorders) | 15
Pain-other (General disorders) | 5
Infection w/o 3-4 neutropenia (Infections and infestations) | 2
Alkaline phosphatase increase (Investigations) | 3
Bilirubin increase (Investigations) | 3
Leukopenia (Investigations) | 19
Lymphopenia (Investigations) | 10
Neutropenia/granulocytopenia (Investigations) | 21
Thrombocytopenia (Investigations) | 14
Anorexia (Metabolism and nutrition disorders) | 2
Dizziness/light headedness (Nervous system disorders) | 7
Headache (Nervous system disorders) | 14
Seizures (Nervous system disorders) | 2
Sensory neuropathy (Nervous system disorders) | 2
Weakness (motor neuropathy) (Nervous system disorders) | 3
Depression (Psychiatric disorders) | 3
Incontinence (Renal and urinary disorders) | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2
Alopecia (Skin and subcutaneous tissue disorders) | 2

LIMITATIONS AND CAVEATS:
Early termination leading to fewer than expected subjects analyzed. With 28 eligible patients estimate of response probability can be estimated to within +/- 19%.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No